CLINICAL TRIAL: NCT04908657
Title: The Effects of Sildenafil for Liver Fibrosis in Adolescents and Adults After Fontan Operation: An Open-label, Randomized Controlled, Pilot Trial.
Brief Title: Sildenafil for Liver Fibrosis in Adolescents and Adults After Fontan Operation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201612207MIPA
Record Dates: First submitted 2017-04-27; First posted 2021-06-01 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Liver Fibrosis
Keywords: Fontan operation; liver fibrosis; sildenafil; treatment
MeSH Terms: conditions — Liver Cirrhosis | interventions — Sildenafil Citrate

STUDY DESIGN:
Intervention Model Description: Open-label, Randomized Controlled
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): treatment group will administrate oral sildenafil 20 mg three times per day for 3 years
  Interventions: Drug: Sildenafil 20 MG
- Control group (No Intervention): the control group will not receive any specific therapy for decreasing the pulmonary vascular resistance

INTERVENTIONS:
Drug: Sildenafil 20 MG — oral sildenafil 20 mg three times per day for 3 years
  Arms: Treatment group

SUMMARY:
Fontan operation is currently the most common procedure performed in patients with single-ventricle physiology. This surgery allows for passive caval blood flow to the pulmonary arteries in the absence of a subpulmonary pump and therefore separating the pulmonary circulation from systemic circulation. However, late hepatic complications such as liver fibrosis, cirrhosis, or even hepatocellular carcinoma are increasingly described in patients with Fontan circulation. The Fontan associated liver disease (FALD) is related to the decreased cardiac output and elevated central venous pressure after Fontan operation. Although the prevalence of FALD is higher than 90% in patients with Fontan circulation. There are no specific medications can reverse the liver fibrosis or prevent the progression of FALD at present. Sildenafil had been used in patients after Fontan operation not only to decrease their pulmonary vascular resistance and central venous pressure, increased systemic cardiac output. Comparing with other oral pulmonary vasodilators, sildenafil is with less possibility of liver toxicity. Therefore, we will conduct a prospective, open-labeled, randomized-controlled study in at least 90 Fontan patients with age > 12 years receiving follow -up at our institute. These patients will be in accordance with the ratio of 1: 1 distribution randomized into two groups, group 1 will receive sildenafil 20 mg three times daily for 3 years and the group will not receive any pulmonary vasodilator as a control. Patients in both group will receive the examinations of liver fibrosis markers, transient ultrasound elastography (FibroScan), diffusion-weighted magnetic resonance imaging (DW-MRI) and cardiopulmonary function test at baseline, 1 year, 2 years and 3 years after initiating treatment. Comparing the results of two groups, we may further clarify the treatment effect of sildenafil on FALD in patients after Fontan procedure.

DETAILED DESCRIPTION:
Research Design and Methods Patients and Methods

1. Study cohort:

   The adolescent and adult patients (age ≥ 12 years) with anatomic and/or functional univentricular heart receive Fontan procedure and are followed at our institute will be included in our study protocol. The expected sample size is 90 candidates, with the ratio of 1:1 distribution randomized into two groups.
2. Inclusion criteria:

   1. Patients age ≥ 12 years with anatomic and/or functional univentricular heart receive Fontan procedure followed at our institute (including the patients with heart failure or pregnancy).
   2. Patients without taking organic nitrates and not allergic to Sildenafil.
3. Exclusion criteria:

   1. The patients cannot safely receive MRI examination, including patients with severe renal dysfunction, or after pacemaker or implantable cardioverter defibrillator implantation.
   2. Patients having known liver disease (such as viral hepatitis, alcoholic liver disease, etc.) other than FALD.
   3. Patients are under sildenafil or any pulmonary vasodilator therapy for lowering pulmonary resistance, or have been using any of these medications in recent 3 months.
4. Methods:

   This is a three-year prospective, open-labeled, randomized-controlled study. After informed consent, eligible patients will be randomly assigned to two groups: the control group will not receive any specific therapy for decreasing the pulmonary vascular resistance, the treatment group will administrate oral sildenafil 20 mg three times per day. The medical records including histories of prior cardiac interventions, hemodynamic data form cardiac catheterization and clinical cardiac performance will be reviewed. Patients who discontinued therapy for any reason will be withdrawn from the trial. All patient will undergo peripheral blood sampling for liver function test, level of circulating biomarkers, acoustic radiation force impulse elastrography and diffusion-weighted magnetic resonance imaging.

   Outcome measures:

   The primary outcome measurement of blood test is the changes from baseline to 1 year, 1.5 years, 2 years, 2.5 years and 3 years in liver fibrosis assessment.

   The measurements include:

   - Liver function tests: including aspartate transaminase (AST) and alanine transaminase (ALT), bilirubin, viral hepatitis markers for hepatitis B and C, gamma-glutamyl transferase (gamma-GT), platelet count, cholesterol, hyaluronic acid, and albumin.

   - Enzyme-linked immunosorbent assay: Serum alfa-macroglobulin, haptoglobin, hyaluronic acid, procollagen type III N-terminal peptide and TIMP metallopeptidase inhibitor 1 levels will be measured with enzyme-linked immunosorbent assay (ELISA) according to manufacturer's instructions (eBioscience, Inc, CA, USA).

   - AST to platelet ratio index (APRI): [{AST (IU/l)/ AST upper limit (IU/l)}× 100]/ platelet count (109/l)

   - Forn's index: 7.811 - 3.131 ln (platelet count (109/L)) + 0.781 ln (gamma-GT (IU/L)) + 3.467 ln (age (y)) - 0.014 (cholesterol (mg/dL))

   - MELD-XI score: 5.11 x ln (total serum bilirubin mg/dL) + 11.76 x ln (serum creatinine mg/dL) + 9.44; serum creatinine and total bilirubin values < 1.0 mg/dL are rounded to 1
   * Transient elastography (TE) TE will be performed using FibroScan (Echosens, France). This machine is equipped with a probe including an ultrasonic transducer mounted on the axis of a vibrator. A vibration transmitted from the vibrator towards the tissue induces an elastic shear wave that propagates through the tissue. These propagations are followed by pulse-echo ultrasound acquisitions and their velocity is measured which is directly related to tissue stiffness. Results are expressed in kilopascal. The examination will be performed on the right lobe of the liver through the intercostal space of the patient. After the area of measurement was located, the examiner pressed the button of the probe to start the acquisition. The measurement depth was between 25 and 65 mm. As suggested by the manufacturer ten successful acquisitions were performed on each patient. Only TE results obtained with 10 valid measurements, with a success-rate of at least 60% and an interquartile range ≤30% were considered reliable. FibroScan failure is defined when less than 10 valid measurements are obtained.
   * Intra-voxel incoherent motion (IVIM) imaging:

   MRI will be performed on a 1.5T MRI system (Magnetom Avanto; Siemens Medical Solution, Erlangen, Germany) with a dedicated, six-channel, torso-array coil. The maximum gradient specificationswere 45 mT/m for amplitude and 200 mT/m/s for the slew rate. The IVIM imaging will be performed in addition to the routine abdomen MRI protocol which included nonenhanced T1-weighted (T1W) and T2-weighted (T2W) imaging, T2W MR cholangiopancreaticography imaging, and contrast-enhanced T1W imaging. Axial IVIM DW images will be acquired using a navigator echo-triggered (PACE [prospective acquisition correction], Siemens) single-shot echo-planar imaging sequence with the following parameters: echo time, 60 ms; repetition time, 2100 ms; echo-planar imaging factor, 115; receiver bandwidth, 1594 Hz per pixel; field of view (FOV), 340 - 256 mm; matrix size, 192 - 115; number of average, 4; section thickness, 7 mm; intersection gap, 1.4 mm; number of sections, 20; and acquisition time, approximately 7 min (variable depending on a patient's respiratory cycle). Instead of bipolar gradients, mono-polar DW gradients which allow for scanning with a shorter echo time, will be used in order to achieve a higher signal-to-noise ratio and to decrease the susceptibility artifacts. An image-based, dynamic distortion correction algorithm will be used to correct for eddy-current-induced distortions. DW gradients (i.e. nine b values of 0, 30, 60, 100, 150, 200, 400, 600, and 900 s/mm2) will be applied in three, orthogonal directions and be subsequently averaged. A k-space-based, parallel imaging technique (generalized auto-calibrating partially parallel acquisition, GRAPPA, Siemens Medical Solutions) will be used with an acceleration factor of 2. Fat suppression will be achieved using a chemical shift-selective, fat-suppression technique.

   The secondary outcome measurement is the changes from baseline to 1 year, 2 years and 3 years in pro-brain natriuretic peptide (NT-pro BNP) levels, New York Heart Association functional classification, 6-minute walk test and cardiopulmonary function test.

   - Methods of cardiopulmonary function test: Equipment The cardiopulmonary exercise test was performed on a cycle ergometer (Ergotest ER 800, Erich Jaeger GmbH & Co., Germany) in an air-conditioned laboratory at a temperature of 22 to 26 oC, barometric pressure of 756 to 772 mmHg, and a relative humidity of 54 to 68%. The blood pressure (TANGO, SunTech Medical Instruments, Inc., North Carolina, USA) and continuous 12-lead electrocardiogram were monitored during test. The expired air was analyzed breath-by-breath using an automatic gas analyzer (Metamax 3B, CORTEX Biophysik GmbH, Leipzig, Germany).

   Exercise Protocol Exercise test was performed at least 2 hours after breakfast. The program began with 2 minutes of data collection in resting on the ergometer, followed by 3 minutes of warm-up cycling with 10 watt, then with load increased by 10 watts per minutes. Patients would exercise as long as they could, and would be stopped based on intolerable dyspnea, fatigue or by supervising physician's safety concerns. Finally, recovery was monitored for more than 3 minutes with unloaded cycling.

   Measurement parameters Exercise cardiopulmonary parameters, including heart rate, 12-lead electrocardiogram, blood pressure, workload (WR), minute ventilation (VE), oxygen consumption (VO2), carbon dioxide production (VCO2), oxygen (O2) pulse, ventilatory equivalent for oxygen (VE/VO2), and ventilatory equivalent for carbon dioxide (VE/VCO2), were processed. The ventilatory threshold (VT) was defined as (1) the VE/VO2 began to increase without a corresponding increase in the VE/VCO2; (2) the end tidal O2 pressure (PO2) began to increase without a decrease in the end tidal CO2 pressure (PCO2); and (3) the VE departed from linearity for VO2.
5. Statistical analysis:

Baseline and demographic characteristics will be summarized by use of means + SDs for continuous variables and percentages for categorical variables. Primary and secondary outcomes changes from baseline will be analyzed by ANCOVA, including terms for treatment group and the baseline variable for the parameter being analyzed. The difference between treatment and control groups is estimated and presented, along with its 2-sided 95% confidence interval and 2-tailed P value.

ELIGIBILITY:
Inclusion Criteria:

1. Patients age ≥ 12 years with anatomic and/or functional univentricular heart receive Fontan procedure followed at our institute (including the patients with heart failure or pregnancy).
2. Patients without taking organic nitrates and not allergic to Sildenafil.

Exclusion Criteria:

1. The patients cannot safely receive MRI examination, including patients with severe renal dysfunction, or after pacemaker or implantable cardioverter defibrillator implantation.
2. Patients having known liver disease (such as viral hepatitis, alcoholic liver disease, etc.) other than FALD.
3. Patients are under sildenafil or any pulmonary vasodilator therapy for lowering pulmonary resistance, or have been using any of these medications in recent 3 months.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-07-03 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Liver MRI | from baseline to 3 years
  Intra-voxel incoherent motion (IVIM) imaging

SECONDARY OUTCOMES:
6-minute walk test | from baseline to 3 years
  6-minute walk test
cardiopulmonary function test | from baseline to 3 years
  Exercise cardiopulmonary parameters
Transient liver elastography | from baseline to 3 years
  Transient liver elastography be performed using FibroScan (Echosens, France)

OTHER OUTCOMES:
pro-brain natriuretic peptide | from baseline to 3 years
  pro-brain natriuretic peptide

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Wei Lu, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- Department of Pediatrics, National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No